CLINICAL TRIAL: NCT01992510
Title: The Effect of Postural Changes on Intraocular Pressure in Silicone Oil-filled Eyes
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Ho Park, Department of Ophthalmology, School of Medicine, Kyungpook National University, Kyungpook National University Hospital
Other Study IDs: KNUH2013
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Silicone Tamponade

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- silicone oil fiiled eye: those with a condition
- fellow eye: the contralateral eye in the same patient

SUMMARY:
The study was conducted to investigate how postural changes including sitting, supine, and LDP(lateral decubitus position) affect the IOP(intraocular pressure) of SO(silicone oil-filled eyes. In addition, this study compared the IOP changes between the SO-filled eyes and the fellow eyes in each body position.

ELIGIBILITY:
Inclusion Criteria:

* patients who had a 23-gauge pars plana vitrectomy
* must be done with SO(silicone oil,5,000 centistrokes) endotamponade using the Accurus system (Alcon Laboratories, Inc, Hünenberg,Switzerland)

Exclusion Criteria:

* previous history or presence of glaucoma or uveitis
* IOP of ≥24 mmHg
* use of any antiglaucoma agents
* narrow angles
* corneal abnormality or diseases that could affect IOP
* refractive error exceeding a spherical equivalent of 6 diopters.

Ages: 33 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: silicone tamponade patients
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Mean IOP(intraocular pressure) at each time point during the change in body position | 100 minutes

SECONDARY OUTCOMES:
IOP(intraocular pressure)differences between the SO(silicone oil)-filled eye and the fellow eyes at each time point during the change in body position | 100 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, School of Medicine, Kyungpook National University, Daegu, Jung-gu, South Korea